CLINICAL TRIAL: NCT02473835
Title: Effects of a Short Term Caloric Restriction on T Cell Activation in Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Unilever R&D (Industry)
Responsible Party: Principal Investigator, Rebecca Travers, Principal Investigator, University of Bath
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UoB - 3 day diet study
Record Dates: First submitted 2015-06-09; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Inflammation
Keywords: T-lymphocyte; Adipose tissue; Inflammation; Calorie restriction
MeSH Terms: conditions — Inflammation | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calorie Restriction (Experimental): Participants reduced calorie intake by 50 % for a period of 3 consecutive days - the target calorie intake for each participant will be determined by a period of energy balance (diet and activity) monitoring.
  Interventions: Other: Calorie restriction; Other: Activity monitoring; Other: Diet monitoring

INTERVENTIONS:
Other: Calorie restriction — Participants will reduce calorie intake by 50 % for a period of 3 consecutive days.
Other: Activity monitoring — For 1 week, participants will be fitted with an activity monitor (Actiheart) to estimate energy expenditure (during the same week as the diet monitoring). The activity and diet monitoring data will be used together to confirm that participants are in a state of energy balance and an average of these 2 values taken - 50 % of this average value will be the target calorie intake for the 3 day calorie restriction period.
Other: Diet monitoring — For 1 week, participants will be asked to record all food and fluids consumed to estimate energy intake (during the same week as the activity monitoring). The activity and diet monitoring data will be used together to confirm that participants are in a state of energy balance and an average of these 2 values taken - 50 % of this average value will be the target calorie intake for the 3 day calorie restriction period.

SUMMARY:
Overweight and obesity are major problems and their complications such as cardiovascular disease and type 2 diabetes mellitus pose great burdens on healthcare systems. There is accumulating evidence to support obesity being a chronic inflammatory disorder mediated in part by the expansion of adipose (fat) tissue.

In addition to adipocytes (fat cells), adipose tissue contains a whole range of other cell types including some immune (white blood) cells. The relative proportions of immune cell subpopulations and interactions between the different cell types within adipose tissue may be important in the development of type 2 diabetes.

Previous research by the investigators has suggested that there may be important differences in the activation status of certain immune cells located in adipose tissue with increased overweight and the production of leptin - an appetite regulating hormone. Properties of adipose tissue and inflammatory cells located within it may therefore be sensitive to changes in our nutritional status.

The purpose of the present study is to investigate changes in T cell activation in adipose tissue alongside other immunometabolic properties before and after a short period of dieting compared to changes in blood.

Participants will include males aged between 35-55 years old who meet the criteria for inclusion. After taking some preliminary measurements and monitoring of normal daily activities, participants will reduce their calorie intake to 50 % of their normal intake/requirements for 3 consecutive days and will attend 1 session of Laboratory testing before and 1 after this period which will take place in the Physiology Laboratories at the University of Bath.

It is hoped that investigating immunometabolic responses within adipose tissue following an acute nutritional challenge will help lead to a better understanding of the development of diseases associated with being overweight and ultimately help in the development of more effective methods for prevention and treatment.

DETAILED DESCRIPTION:
The aim of this research is to investigate whether the immunometabolic properties of adipose tissue and the inflammatory cells located within it can be modified by short term changes in nutritional status.

Following advertisement of the study, interested potential participants will be asked to contact the Chief Investigator for further information via email/telephone correspondence. There will be an initial assessment of eligibility based on inclusion/exclusion criteria and, if these requirements are met, the potential participant will be invited to a meeting to further discuss the trial. After they have read the participant information sheet and seen the flowchart outlining the timeline for the study, if they would like to take part, they will be asked to sign a consent form. Dates will then be scheduled for some preliminary anthropometric measurements, 1 week of diet and physical activity monitoring and 3 days of calorie restriction with trial dates either side.

Preliminary measurements:

Preliminary testing will include anthropometric measurements of height, weight, waist and hip circumferences, sagittal waist height and blood pressure. Participants will also have their body composition precisely assessed using a dual energy X-ray absorptiometer (DEXA). These measurements will take place at the University of Bath Physiology Laboratories.

Monitoring of energy balance:

For 1 week, participants will be fitted with a physical activity monitor (Actiheart™) and asked to record a corresponding diary of their physical activity during this period to aid its interpretation and allow a more accurate calculation of average daily activity energy expenditure. Participants will also be asked to record their food and drink intake during this period so their corresponding energy intake during this period can be analysed and thus their 'energy balance' can be estimated. Participants should not make any conscious changes to their normal lifestyle habits/routines during this period. This analysis will then be used to write a 'diet prescription' for the 3 days to ensure the participant will receive 50 % of their 'normal' calorie intake using foods they would normally consume.

Main trial day 1:

In the 2 days prior to the first main trial day, participants should refrain from performing any strenuous physical activity. In the 24 hours prior, participants should also refrain from consuming any alcohol or caffeine. Participants should arrive at the Physiology Resting Laboratory in the morning following a 10 hour fast (approximately 8 am) where blood pressure will be measured and a saliva sample collected. A cannula will be inserted into a forearm vein and baseline blood sample(s) taken for analysis of metabolic/inflammatory markers and isolation of T cells. A fat sample will also be obtained using a needle aspiration technique. The participant will then be asked to consume a glucose drink consisting of 75 g anhydrous glucose (113 mL Polycal and 87 mL of water) and a cannula blood sample taken every 15 minutes for the following 2 hours.

Intervention - 3 day calorie restriction:

For the following 3 days, participants will be instructed to consume a diet calculated to be 50% of their 'normal' energy intake by reducing the proportions of the normal diet consumed. No strenuous physical activity should be performed by the participant for the last 2 days of this 3 day period and on the final day of this intervention, no caffeine or alcohol should be consumed.

Main trial day 2:

The following day after the 3 days of calorie restriction, participants will arrive at the laboratory at the same time as on main trial day 1 (to minimise variation in timing of sample collection) and will undergo exactly the same procedures.

Analysis:

On the day of the trial whole blood will be analysed for white blood cell count. Plasma and serum samples will be extracted from the whole blood via centrifugation and stored at -80 degrees C. Monocytes and T lymphocytes (populations of white blood cells) will also be isolated from whole blood and stored to later assess changes in their proportions and activation following the calorie restriction period. In each fat sample, separate portions of either adipose tissue or adipocytes (isolated from the other cells within the adipose tissue using a digestion method) will be cultured and media collected for later investigations. The remaining cells from the adipose tissue (SVF) will also be stored for later analysis of cell populations and their activation using flow cytometry, and expression/secretion analysis. mRNA expression will also be examined in adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference > 94 cm
* Weight stable for more than 3 months (no change in weight +/- 3 %)
* Non-smoker

Exclusion Criteria:

* Personal history of/existing cardiovascular disease, metabolic disease or dyslipidaemia
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in T cell activation in adipose tissue in response to calorie restriction | 3 days
  T-lymphocytes will be isolated from adipose tissue samples taken before and after 3 days of 50 % calorie restriction and levels of their activation will be assessed by flow cytometry.

SECONDARY OUTCOMES:
Changes in T cell activation in blood in response to calorie restriction | 3 days
  T-lymphocytes will be isolated from blood samples taken before and after 3 days of 50 % calorie restriction and levels of their activation will be assessed by flow cytometry.
Changes in IL-6 mRNA expression by adipose tissue | 3 days
  mRNA expression of IL6 will be measured in adipose tissue samples obtained before and after 3 days of 50 % calorie restriction to assess for inflammatory changes in adipose tissue.
Changes in IL-6 secretion by adipose tissue | 3 days
  Adipose tissue explants will be cultured for 3 hours using samples obtained before and after 3 days of 50 % calorie restriction to assess for changes in IL-6 secretion.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Thompson, PhD, Principal Investigator — Professor
Locations (1):
- University of Bath - Department for Health, Bath, Bath and North East Somerset, United Kingdom

REFERENCES:
- [Background] Travers RL, Motta AC, Betts JA, Bouloumie A, Thompson D. The impact of adiposity on adipose tissue-resident lymphocyte activation in humans. Int J Obes (Lond). 2015 May;39(5):762-9. doi: 10.1038/ijo.2014.195. Epub 2014 Nov 12. PMID 25388403